CLINICAL TRIAL: NCT01954290
Title: Treatment of Brain Edema and Herniation Secondary to Ischemic or Hemorrhagic Stroke
Brief Title: Study of Stroke Related Edema Treatments
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator is leaving the institution.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 136-2013
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Acute Cerebrovascular Accident; Cerebral Edema
Keywords: Stroke; Brain Edema; Brain Herniation; Conivaptan
MeSH Terms: conditions — Stroke; Brain Edema | interventions — conivaptan; Saline Solution, Hypertonic; Sodium Chloride; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertonic Saline (3%) and/or Mannitol arm (Active Comparator): The subjects in this arm will be given hypertonic saline and/or Mannitol.
  For hypertonic saline,various concentrations are used clinically,up to 30-mL boluses of 23.4% saline.Rapid increases in sodium in this context do not appear to cause other neurologic complications observed with rapid correction of hyponatremia.Sodium levels up to 160 mmol/L may be acceptable,beyond which it may lead to worsening delirium,seizures,and overall poor outcome.
  For Mannitol,every 4 hours serum osmolarity,serum glucose,urea,sodium and potassium will be measured till the therapy is given.Major complications include hypovolemia and hypotension.Strict fluid goals and volume replacement are essential.Impaired mannitol clearance may manifest as nephrotoxicity.Common practice includes repeating measurements of serum osmolarity and withholding repeat doses of mannitol when osmolarity exceeds 320 milliosmol(mOsm).Monitoring the osmole gap may be a more sensitive method for discerning mannitol clearance.
  Interventions: Drug: Hypertonic saline; Drug: Mannitol
- Conivaptan arm (Experimental): The subjects in this arm will be given infusion of Conivaptan.
  Interventions: Drug: Conivaptan

INTERVENTIONS:
Drug: Conivaptan — Intravenous conivaptan 20 mg infused over 30 minutes as a loading dose, followed by a continuous infusion of 20 mg over 24 hours (0.83 mg/hour) for 2-4 days; may increase to a maximum dose of 40 mg over 24 hours (1.7 mg/hour) if serum sodium is not rising sufficiently; total duration of therapy not to exceed 4 days.
  Other Names: Vaprisol
  Arms: Conivaptan arm
Drug: Hypertonic saline — Hypertonic saline in the dose of 30ml/hr, with every 4 hourly measurements of serum osmolarity, serum sodium and potassium. Hypertonic saline will be increased by 30 ml to achieve target serum sodium of 150-160 and serum osmolarity 300-320
  Other Names: Sodium chloride injection (3% or 5%); Brand name: Viaflex
  Arms: Hypertonic Saline (3%) and/or Mannitol arm
Drug: Mannitol — Mannitol given at the dose of 0.5 to 1.0 gm/kg IV over 10-20 minutes. Maximum effect is seen in 20 minutes and duration of action is 4 hours. Repeat doses of 0.25 to 0.5 gm/kg Q 4-6 hours are normally frequently used.
  Other Names: Brand name: Osmitrol
  Arms: Hypertonic Saline (3%) and/or Mannitol arm

SUMMARY:
Stroke remains the fourth leading cause of death in the United States (second worldwide) and a leading cause of long-term disability, resulting in total direct and indirect costs of approximately $73.7 billion annually. The failure of novel therapies in clinical trials demonstrates that the complex neural response to stroke must be targeted at multiple levels to improve patient outcomes. Despite significant improvements in stroke treatment and management, 1 year survival rate among stroke patients aged 65 years or more is around 25%, and 5- year survival rate amounts to approximately 50%. The highest chances of death are within 30 days of stroke. Mortality increases due to worsening brain dysfunction, elevated intracranial pressure (ICP), and other comorbid conditions.

Treatments aimed at reducing post-stroke cytotoxic edema may reduce the risk for development of malignant stroke and mortality. Current treatments such as osmo-therapy and hemicraniectomy have substantial limitations, and mortality remains high, despite these measures outcomes remain unsatisfactory. There is a great need for alternative medical approaches which are safe, predictable, and help to ameliorate post stroke edema.

DETAILED DESCRIPTION:
Previous work has demonstrated the pathophysiological role of arginine-vasopressin (AVP) in ischemic stroke. The mechanism of action of AVP is by 3 receptor subtypes: V1a, V1b and V2 expressed in brain, pituitary gland, myocardium, vasculature and kidneys. The role of the vasopressin receptors V1a and or V2 subtype in cerebral edema formation after ischemic stroke remains controversial. The V1a receptor antagonism causes platelet inhibition, aquaporin-4 up regulation; reduce infarct size and vasodilation. V1 antagonists has also been shown to prevent ischemia-induced cerebral edema development, suggesting that the V1 vasopressin receptor is important in water regulation in brain cells. Another study indicated that the vasopressin receptor V1 is involved in the pathogenesis of secondary brain damage after focal cerebral ischemia. Recently, few studies have demonstrated that a V2 receptor antagonist (OPC-31260), may be one of the effective drugs for the early treatment of cytotoxic edema and brain injury. Treatment of OPC-31260 ameliorated cerebral neurological deficit in transgenic (GET-1) mice after water intoxication. Treatment of OPC-31260 also significantly abolished water accumulation and down regulated Aquaporin-4 (AQP-4) expression level in GET-1 mice after water intoxication. The intensity of AQP-4 staining was almost comparable with that of the controls without water intoxication. It was also shown that OPC-31260 at doses of 10 to 30 mg/kg produced a dose-dependent inhibition of subarachnoid hemorrhage-induced cerebral edema formation, accompanied by an increase in urinary volume and decrease in urine osmolality without a significant alteration of urine electrolytes. OPC-31260 is also effective in treating water retention diseases, such as hyponatremia caused by inappropriate antidiuretic hormone secretion, congestive heart failure, and liver cirrhosis. V2 receptor antagonism will also help in abolishing water accumulation, decreased Glial Fibrillary Acidic Protein (GFAP) in astrocytes and most importantly causes renal tubule-selective diuretic effect called aquaresis (electrolyte sparing diuresis), which may have additional benefit in the reduction of cerebral edema.

This combined approach of V1a and V2 AVP receptor antagonism will lead to attenuation of ischemia related cerebral edema and infarct volume by modulating ischemia-evoked AQP-4 expression. This effect should help behavior and mortality which in turn will improve outcome in stroke patients. The purpose of this project is to test the effect of the mixed V1a and V2 receptor blockade on ischemic or hemorrhagic stroke outcome.

In summary, the investigators are using the approach of mixed vasopressin antagonism on post stroke edema, infarct volume and outcome. This research will lead to a greater understanding of the roles and interactions of the different AVP receptors and pathophysiology of post stroke cytotoxic edema. New information on the effects of mixed blockade of V1a and V2 receptors on the prevention of cytotoxic edema post stroke will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age ≥18 years and ≤80 years at the time of screening.
* Hemorrhagic stroke or large vessel ischemic stroke patients diagnosed by MRI or CT scan of Head.
* Subjects who have presented to hospital within 24 hours of symptom onset.
* The subject or his/ her legal representative is willing to undergo informed consent process prior to enrollment into this study.

Exclusion Criteria:

* Subject with age < 18 years and >80 years at the time of screening.
* Subjects with absence of stroke by imaging of brain by CT scan or MRI.
* Lacunar stroke or small vessel stroke.
* Time of symptom onset cannot be determined.
* Subjects with renal or hepatic failure.
* Subjects with hypovolemia or hypotension as determined by the study team.
* Subjects with hypernatremia.
* Subject who is pregnant or lactating.
* Subject is already participating in other investigational clinical trial.
* The subject or legal representative is unable to provide informed consent.
* The subject is medically unstable to participate in the trial as determined by the principal investigator.
* The subject has any end stage medical condition as determined by the principal investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Score | At the time of discharge from hospital, and 3 months after initial event
  The modified Rankin Scale (m-RS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people after they have suffered a stroke.It is one of the most widely used clinical outcome measure for stroke clinical trials. The score is given according to following scale.
  0- No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
National Institutes of Health Stroke Severity (NIHSS) scale | At the time of discharge from hospital, and 3 months after initial event
  NIHSS is a tool used by healthcare providers to objectively quantify the degree of impairment caused by a stroke. It is composed of 11 items. Each item scores a specific ability between a score of 0-4. Usually, for each item, a score of 0 indicates normal function in that specific ability, while a higher score indicates some level of impairment. The individual scores from each item are added together to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Neurological status of the subject | At the time of discharge from hospital, and 3 months after discharge
  Neurological status of a stroke subject is assessed by physical neurological examination of the subject by a qualified neurologist. It is one of the most important aspect in determining neurological health of a subject after treatment for stroke. It also helps to determine stroke severity and prognosis.

SECONDARY OUTCOMES:
All cause mortality data | 3 months after initial event
  Mortality data indicates the severity of stroke.

OTHER OUTCOMES:
MRI brain- findings | 3 Months after Initial Event
  MRI of the Brain.

CONTACTS AND LOCATIONS:
Overall Officials: Vishnumurthy Shushuthra Hedna, MD, Principal Investigator — University of Florida; Michael F Waters, MD, Study Director — University of Florida